CLINICAL TRIAL: NCT03426969
Title: A Pilot Study of Reduced Intensity HLA-Haploidentical Hematopoietic Cell Transplantation With Post-Transplant Cyclophosphamide in Patients With Advanced Myelofibrosis
Brief Title: Combination Chemotherapy, Total Body Irradiation, and Donor Blood Stem Cell Transplant in Treating Patients With Primary or Secondary Myelofibrosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0375; NCI-2018-00910 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0375 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2018-02-02; First posted 2018-02-08 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Primary Myelofibrosis; Secondary Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor; fludarabine phosphate; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Melphalan; Mycophenolic Acid; Tacrolimus; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (combination chemotherapy, TBI, HCT) (Experimental): Patients receive melphalan IV over 30 minutes on days -5, fludarabine phosphate IV over 1 hour on days -5 to -2. Patients undergo TBI on day -1 and HCT on day 0. Patients then receive cyclophosphamide IV over 1-2 hours on days 3 and 4. Beginning on day 5, patients receive tacrolimus IV continuously for approximately 2 weeks, then PO for 6 months followed by a taper, mycophenolate mofetil PO TID until day 100, and filgrastim SC daily from day 7 until continued until ANC > 1,500/mm^3 for 3 consecutive days. Treatment continues in the absence of disease progression or unexpected toxicity.
  Interventions: Drug: Cyclophosphamide; Biological: Filgrastim; Drug: Fludarabine Phosphate; Procedure: Hematopoietic Cell Transplantation; Drug: Melphalan; Drug: Mycophenolate Mofetil; Drug: Tacrolimus; Radiation: Total-Body Irradiation

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Biological: Filgrastim — Given SC
  Other Names: G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Procedure: Hematopoietic Cell Transplantation — Undergo HCT
  Other Names: HCT; Hematopoietic Stem Cell Transplantation; HSCT; Stem Cell Transplant; stem cell transplantation
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine nitrogen mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Drug: Tacrolimus — IV or PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TBI; TOTAL BODY IRRADIATION; Whole Body Irradiation; Whole-Body Irradiation

SUMMARY:
This early phase I trial studies the side effects of combination chemotherapy, total body irradiation, and donor blood stem cell transplant in treating patients with primary or secondary myelofibrosis. Drugs used in chemotherapy, such as melphalan, fludarabine phosphate, cyclophosphamide, tacrolimus, mycophenolate mofetil, and filgrastim work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays to kill cancer cells and shrink tumors. Giving combination chemotherapy and total body irradiation before a donor blood stem cell transplant helps to stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and tolerability of reduced-intensity (FM) haploidentical hematopoietic cell transplantation (Haplo-HCT) followed by post-transplant cyclophosphamide (PTCy) in patients with advanced myelofibrosis (MF), as assessed by the evaluation of toxicities, including type, frequency, severity, attribution, time course and duration.

SECONDARY OBJECTIVES:

I. To summarize and evaluate hematologic (neutrophil and platelet) recovery. II. To estimate graft failure-free survival (GFS) at 100-days post-transplant. III. To estimate overall survival (OS), progression-free survival (PFS) and cumulative incidence (CI) of relapse/progression, and non-relapse mortality (NRM) at 100-days, 1-year, and 2-year post transplant.

IV. To estimate the cumulative incidence of acute graft-versus-host disease (GvHD), grade II-IV, at 100-days post-transplant (per Keystone Consensus modification of the Glucksberg criteria).

V. To estimate the cumulative incidence of chronic GvHD at 1-year and 2-year post transplant (per National Institute of Health [NIH] Consensus Criteria).

VI. To characterize the severity and extent of acute and chronic GvHD.

OUTLINE:

Patients receive melphalan intravenously (IV) over 30 minutes on days -5, fludarabine phosphate IV over 1 hour on days -5 to -2. Patients undergo total body irradiation (TBI) on day -1 and hematopoietic stem cell transplant (HCT) on day 0. Patients then receive cyclophosphamide IV over 1-2 hours on days 3 and 4. Beginning on day 5, patients receive tacrolimus IV continuously for approximately 2 weeks, then orally (PO) for 6 months followed by a taper, mycophenolate mofetil PO thrice daily (TID) until day 100, and filgrastim subcutaneously (SC) daily from day 7 until continued until absolute neutrophil count (ANC) > 1,500/mm^3 for 3 consecutive days. Treatment continues in the absence of disease progression or unexpected toxicity.

After completion of study treatment, patients are followed up at 1, 3, 6, 9, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary or secondary Myelofibrosis with transplant indication by DIPSS-plus (> intermediate -1);
* Age 18-70; patients >/= age 50 must have an comorbidity score (HCT-CI) </= 4 (Sorror). The Principal Investigator is the final arbiter for comorbidity;
* Patients can be in chronic phase (CP) with BM blast count </= 10% or after progression to AML and achieved </= 5% BM blasts (morphologic CR prior to transplant);
* Lack of an HLA matched donor or need to proceed fast to transplantation when a patient does not have an immediately available matched unrelated donor (typed by high-resolution in the registry);
* Performance status >/=70% (Karnofsky); patients > 50 years should have adequate cognitive function; any concerns regarding cognitive function should be addressed by a Geriatrician/Neurologist;
* Adequate organ function: ALT/AST/billirubin </= 5X UNL, creatinine clearance > 50mls/min (calculated with Cockroft-Gault formula); LVEF >/= 50%, DLCOc >/= 50%;
* Prior treatment with JAK2 inhibitor therapy is not excluded. Patients on a JAK2 inhibitor may continue through conditioning until Day -3 then tapered at the discretion of the investigator.

Exclusion:

* Evidence of portal hypertension with varices, ascites, or hepatic encephalopathy;

  ->10% bone marrow blasts at transplant if no history of AML and >5% if had previous progression to AML;
* HIV positive; active hepatitis B or C;
* Patients with active infections. The PI is the final arbiter of the eligibility;
* Liver cirrhosis;
* Prior CNS involvement by tumor cells;
* Severe pulmonary hypertension (PHT) (On echo or right side cardiac catheterization);
* History of another primary malignancy that has not been in remission for at least 3 years (the following are exempt from the 3-year limit: non-melanoma skin cancer, fully excised melanoma in situ [Stage 0], curatively treated localized prostate cancer, and cervical or breast carcinoma in situ on biopsy or a squamous intraepithelial lesion on PAP smear);
* Positive Beta HCG test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization;
* Noncompliance - Inability or unwillingness to comply with medical recommendations regarding therapy or follow-up, including smoking tobacco. Smoking cessation is a standard teaching practice prior to admission for all patients undergoing stem cell transplant. Any patient who refuses to stop smoking prior to transplant will not be eligible for this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-09-21 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to day +100 post-hematopoietic cell transplantation (HCT)
  Observed toxicities will be tabulated and summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study regimen and reversibility or outcome.

SECONDARY OUTCOMES:
Overall survival | Up to 24 months
  Estimated will be calculated using the Kaplan-Meier product-limit method. Distributions will be compared using the log-rank test. Cox proportional hazards regression will be used to assess the association between survival endpoints and clinical and disease covariates of interest.
Progression-free survival | Up to 24 months
  Estimated will be calculated using the Kaplan-Meier product-limit method. Distributions will be compared using the log-rank test. Cox proportional hazards regression will be used to assess the association between survival endpoints and clinical and disease covariates of interest.
Graft failure-free survival | Up to 24 months
  Estimates will be calculated using the Kaplan-Meier product-limit method. Distributions will be compared using the log-rank test. Cox proportional hazards regression will be used to assess the association between survival endpoints and clinical and disease covariates of interest.
Time to neutrophil recovery | Up to 24 months
  Will be estimated using the Kaplan-Meier product-limit method. Distributions will be compared using the log-rank test. Cox proportional hazards regression will be used to assess the association between survival endpoints and clinical and disease covariates of interest.
Time to platelet recovery | Up to 24 months
  Will be estimated using the Kaplan-Meier product-limit method. Distributions will be compared using the log-rank test. Cox proportional hazards regression will be used to assess the association between survival endpoints and clinical and disease covariates of interest.
Non-relapse mortality (NRM) | Up to 24 months
  The cumulative incidence of relapse/progression with a competing risk of NRM will be estimated in a competing risks framework. Analyses to assess the association between the cumulative incidence of the above parameters and clinical and disease covariates of interest will be performed using the method of Fine and Gray.
Acute graft versus host disease (GvHD) | Up to 24 months
  Will be estimated in a competing risks framework with competing risks of relapse and NRM. Analyses to assess the association between the cumulative incidence of the above parameters and clinical and disease covariates of interest will be performed using the method of Fine and Gray.
Chronic GvHD | Up to 24 months
  Will be estimated in a competing risks framework with competing risks of relapse and NRM. Analyses to assess the association between the cumulative incidence of the above parameters and clinical and disease covariates of interest will be performed using the method of Fine and Gray.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan O Ciurea, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org